CLINICAL TRIAL: NCT01603095
Title: A Multicenter, Multinational Clinical Assessment Study for Pediatric Patients With Achondroplasia
Status: Completed | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 111-901; 2017-000701-21 (EudraCT Number)
Record Dates: First submitted 2012-05-11; First posted 2012-05-22 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Achondroplasia
Keywords: Achondroplasia; dwarfism
MeSH Terms: conditions — Achondroplasia; Dwarfism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Growth measurements: Approximately 500 patients will be enrolled. Patients from birth to <= 17 years on the date of consent will be enrolled. Approximately equal numbers of boys and girls will be enrolled.

SUMMARY:
Multicenter, multinational study to collect consistent baseline growth measurements on pediatric patients with Achondroplasia being considered for subsequent enrollment in future studies sponsored by BioMarin. No study drug is administered.

ELIGIBILITY:
Inclusion Criteria:

* Parent(s) or guardian(s) willing and able to provide signed informed consent after the nature of the study has been explained and prior to performance of any research-related procedure. Also, willing and able to provide written assent (as needed) after the nature of the study has been explained and prior to performance of any research-related procedure.
* Aged 0 to <= 17 years, inclusive, at study entry.
* Have ACH, documented by clinical diagnosis
* Are ambulatory and able to stand without assistance (not applicable for infants)
* Are willing and able to perform all study procedures as physically possible.

Exclusion Criteria:

* Have hypochondroplasia or short stature condition other than ACH (e.g., trisomy 21, pseudoachondroplasia)
* Have any of the following disorders:

  * Hypothyroidism
  * Insulin-requiring diabetes mellitus
  * Autoimmune inflammatory disease
  * Inflammatory bowel disease
  * Autonomic neuropathy
* Have an unstable clinical condition likely to lead to intervention during the course of the study, including progressive cervical medullary compression
* Growth plates have fused
* Have a history of any of the following:

  * Renal insufficiency
  * Anemia
* Cardiac or vascular disease, including the following:

  * Cardiac dysfunction (abnormal echocardiogram [ECHO] including left ventricle [LV] mass) at Screening Visit
  * Hypertrophic cardiomyopathy
  * Congenital heart disease
  * Cerebrovascular disease, aortic insufficiency
  * Clinically significant atrial or ventricular arrhythmias
* Current treatment with antihypertensive medications angiotensin-converting enzyme (ACE) inhibitors, angiotensin II receptor blockers, diuretics, beta-blockers, calcium-channel blockers, cardiac glycosides, systemic anticholinergic agents, any medication that may impair or enhance compensatory tachycardia, drugs known to alter renal function that is expected to continue for the duration of the study
* Have been treated with growth hormone, insulin-like growth factor 1 (IGF-1), or anabolic steroids in the previous 6 months or long-term treatment (> 3 months) at any time
* Have had regular long-term treatment (> 1 month) with oral corticosteroids (low-dose ongoing inhaled steroid for asthma is acceptable)
* Concomitant medication that prolongs the QT/QTc interval within 14 days or 5 half-lives, whichever is longer, before the Screening visit
* Have used any other investigational product or investigational medical device for the treatment of ACH or short stature
* Have had bone-related surgery or expected to have bone-related surgery during the study period. Subjects with previous limb-lengthening surgery may enroll if surgery occurred at least 18 months prior to the study and healing is complete without sequelae.
* Have any condition that, in the view of the Investigator, places the patient at high risk of poor compliance with the visit schedule or of not completing the study.
* Concurrent disease or condition that, in the view of the Investigator, would interfere with study participation

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Approximately 500 patients will be enrolled. Patients from birth to <= 17 years, inclusive, on the date of consent will be enrolled. Approximately equal numbers of boys and girls will be enrolled.
Sampling Method: Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2012-04; Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Collection of consistent growth measurements | Assessed every 3 months for up to 84 months
  Patients will be screened and undergo a series of growth measurements on Day 1 and every 3 months thereafter. No study drug is administered.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (20):
- United States (9):
  - Harbor-UCLA Medical Center, Los Angeles, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Emory University, Decatur, Georgia
  - Ann and Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin, Children's Hospital, Milwaukee, Wisconsin
- Australia (2):
  - Murdoch Children's Research Institute, Parkville, Victoria
  - The Children's Hospital at Westmead, Westmead
- Japan (3):
  - Osaka University Hospital, Osaka
  - Saitama Children's Medical Center, Saitama
  - Tokushima University Hospital, Tokushima
- Spain (3):
  - Institut Catala de Traumatologica I Medicina de l'Esport, Barcelona
  - Hospital Sant Joan de Deu Barcelona, Barcelona
  - Hospital Universitario Virgen de la Victoria, Málaga
- Acibadem University School of Medicine, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - Guy's and St. Thomas NHS Foundation Trust Evelina Children's Hospital, London
  - Sheffield Children's NHS Foundation Trust, Sheffield

REFERENCES:
- [Derived] Savarirayan R, Irving M, Harmatz P, Delgado B, Wilcox WR, Philips J, Owen N, Bacino CA, Tofts L, Charrow J, Polgreen LE, Hoover-Fong J, Arundel P, Ginebreda I, Saal HM, Basel D, Font RU, Ozono K, Bober MB, Cormier-Daire V, Le Quan Sang KH, Baujat G, Alanay Y, Rutsch F, Hoernschemeyer D, Mohnike K, Mochizuki H, Tajima A, Kotani Y, Weaver DD, White KK, Army C, Larrimore K, Gregg K, Jeha G, Milligan C, Fisheleva E, Huntsman-Labed A, Day J. Growth parameters in children with achondroplasia: A 7-year, prospective, multinational, observational study. Genet Med. 2022 Dec;24(12):2444-2452. doi: 10.1016/j.gim.2022.08.015. Epub 2022 Sep 16. PMID 36107167
- [Derived] Chan ML, Qi Y, Larimore K, Cherukuri A, Seid L, Jayaram K, Jeha G, Fisheleva E, Day J, Huntsman-Labed A, Savarirayan R, Irving M, Bacino CA, Hoover-Fong J, Ozono K, Mohnike K, Wilcox WR, Horton WA, Henshaw J. Pharmacokinetics and Exposure-Response of Vosoritide in Children with Achondroplasia. Clin Pharmacokinet. 2022 Feb;61(2):263-280. doi: 10.1007/s40262-021-01059-1. Epub 2021 Aug 25. PMID 34431071
- [Derived] Savarirayan R, Irving M, Bacino CA, Bostwick B, Charrow J, Cormier-Daire V, Le Quan Sang KH, Dickson P, Harmatz P, Phillips J, Owen N, Cherukuri A, Jayaram K, Jeha GS, Larimore K, Chan ML, Huntsman Labed A, Day J, Hoover-Fong J. C-Type Natriuretic Peptide Analogue Therapy in Children with Achondroplasia. N Engl J Med. 2019 Jul 4;381(1):25-35. doi: 10.1056/NEJMoa1813446. Epub 2019 Jun 18. PMID 31269546